CLINICAL TRIAL: NCT05766657
Title: Evaluation of the Effect of an Anti-inflammatory Diet Built on the Basis of the Gut Microbiota in Children with Type 1 Diabetes and Obesity
Brief Title: Evaluation of an Anti-inflammatory Diet in Autoimmune and Metabolic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Marika Falcone, Principal Investigator, IRCCS San Raffaele
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUTRI-DIET
Record Dates: First submitted 2022-12-02; First posted 2023-03-13 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Type1 Diabetes; Obesity
Keywords: Gut microbiome; Inflammation; Type 1 Diabetes; Obesity; Immunology; Gut barrier; Intestinal barrier; Extra-intestinal diseases
MeSH Terms: conditions — Obesity; Inflammation; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomized, multicenter, 2-arm, parallel-group, single-blind controlled clinical trial (1:1 allocation ratio)
Who Masked: Participant, Care Provider
Masking Description: Single blind: Apart from clinical nutritionists who will be involved in dietary counseling, physicians and all project staff who will be responsible for patient selection and follow-up, along with biostatisticians, will be blinded to the intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Children with obesity or T1D will be randomized into this group. An individualized dietary approach will be used in this group of children.
  Interventions: Dietary Supplement: Microbiome-targeted diet
- Control Group (Placebo Comparator): children assigned to the control group will receive generic advice based on European dietary guidelines for obesity or follow their usual diet in the case of children with T1D.
  Interventions: Dietary Supplement: Usual care diet

INTERVENTIONS:
Dietary Supplement: Microbiome-targeted diet — The gut microbiota (on stool) and metabolic profile (on stool and urine) will be analyzed at time 0, and the dietary plan will contain specific directions aimed at restoring a proper metagenomic and metabolomic profile of the microbiota.
  Arms: Intervention group
Dietary Supplement: Usual care diet — Subjects on the control group will receive general dietetic advice for Obesity or T1D
  Arms: Control Group

SUMMARY:
The overall objective of the study is to provide personalized nutritional advice based on the gut microbiota profile of children with type 1 diabetes (T1D) or obesity.

Specifically, the primary objective of NUTRI-DIET is to validate a dietary model aimed at restoring bacterial species and/or anti-inflammatory metabolites in order to prevent extra-intestinal diseases characterized by dysbiosis, such as T1D and obesity.

The primary endpoints of the study will be to monitor the glycemic control indices, i.e., blood glucose (mean of glycemic values, percentage of time-in-range value (TIR), which will be displayed by glycemic sensor) and glycated hemoglobin for diabetic children and Body mass index (BMI) z-score according to World Health Organization (WHO) recommendations (WHO BMI-for-age boys; WHO BMI-for-age girls) for obese children.

The secondary objective of the study is to characterize the microbiota profile of the study patients and to test the algorithm under development built from the integration of diet and and gut microbiota composition data that were obtained during the previous observational study NUTRI-T1D.

DETAILED DESCRIPTION:
Randomized, multicenter, 2-arm, parallel-group, single-blind controlled clinical trial (1:1 allocation ratio) with 1 group of patients with obesity (N=20) or type 1 (n=20) treated with standard obesity treatment diet or usual diet (diabetic children) and 1 group (N=20 for obesity and (N=20 for type 1 diabetes) treated with the same diets to which nutritional advice derived from microbiota analysis (NUTRI-DIET) will be added.

The study will last 12 months with an intervention phase (personalized diet) lasting 3 months.

The research includes an enrollment phase that may extend up to 9 months depending on the number of patients enrolled. The enrollment phase will be considered finished once a total of 80 patients (i.e., 40 pediatric patients with type 1 diabetes and 40 obese pediatric patients) are enrolled. During the patient enrollment phase, relevant clinical information (biological samples as faeces, urines and blood and questionnaires on diet habits, physical activity and stress) will be collected concurrently. Tests will be performed once enrollment is completed on samples from all patients collected at the time of enrollment (microbiota analysis on stool, metabolome analysis on stool and urine, serological gut barrier markers analysis on serum). Obese and/or diabetic children will be randomized to the intervention or control group. Randomization will be done according to age (≤12: >12), gender and pathology (diabetes or obesity).

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for participation will be children diagnosed with obesity (BMI > 95th percentile) and type 1 diabetes aged 8-18 years
2. Signature of informed consent

Exclusion Criteria:

1. Children with any acute or chronic disease (cancer, infection, other), gastrointestinal disease, cardiovascular disease, chronic kidney disease, parathyroid disease, diseases requiring regular phlebotomies, and other chronic diseases that could affect the results of the present study
2. Taking medications other than insulin, including hypolipidemic and antihypertensive drugs
3. Use of medications that could affect the results of the study, including systemic glucocorticoids and antibiotics (in the three months prior to the study)
4. Recent weight loss or weight gain (> 3 kg), (in the 3 months preceding the study)
5. Blood transfusion in the last 3 months prior to blood sampling
6. Use of dietary supplements, including multivitamins, fish oil capsules, minerals and trace elements (three months prior to and throughout the study period)
7. Inability (physically or psychologically) to comply with the procedures required by the protocol
8. Children with specific eating disorders, which may hinder the research results

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Glycemia | Up to 3 months
  Blood glucose levels (mg/dL) will be measured in diabetic children.
Glycemic control by glycated hemoglobin (HbA1c) monitoring | Up to 3 months
  The percentage of glycated hemoglobin (HbA1c, %) in the blood will be measured in diabetic children.
Glycemic control by Time-in-Range (TIR) monitoring | Up to 3 months
  TIR values - that is the percentage of time in which blood glucose (blood sugar) remains in the safe target range of 70-180mg/dL - will be monitored in diabetic children by extracting the recorded data from the continuous glucose monitoring (CGM) device (sensor).
Body mass index (BMI) | Up to 3 months
  The BMI z-score in obese children will be measured, according to WHO recommendations (WHO BMI-for-age boys; WHO BMI-for-age girls).

SECONDARY OUTCOMES:
Metagenomic analysis | Up to 3 months
  Changes in gut microbiota composition following personalized microbiome-targeted diet, as assessed by 16S ribosomal RNA (rRNA) sequencing on DNA extracted from patient-derived fecal samples.
Metabolomic analysis | Up to 3 months
  Changes in microbiota-derived metabolites following personalized microbiome-targeted diet, as assessed by Mass Spectrometry on patient-derived fecal and urine samples.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Pediatric Unit, Milan, Milano
  - Autoimmune Pathogenesis Unit, Milan, Milan

IPD SHARING:
Plan to Share IPD: No